CLINICAL TRIAL: NCT01672944
Title: Evaluating Biobanking Educational Tools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MCC-16448
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Neoplasm
Keywords: Biological specimen banks; Health education; Tissue banks; Health care survey; Tissue
MeSH Terms: conditions — Neoplasms; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TBCCN-developed educational materials (Experimental): Biobanking educational DVD and booklet kit developed by the Tampa Bay Community Network (TBCCN) Center. English kit is entitled "Biobanking Hope for a Cancer Cure", and Spanish kit is entitled "Biobanco: Una esperanza de cura para el cancer."
  Interventions: Other: TBCCN-developed educational materials
- Control Group (Other): Biobanking educational Brochure developed by the National Cancer Institute. English brochure is entitled "Providing your Tissue for Research: What you need to Know", Spanish brochure is entitled "Lo que usted debe saber antes de dar sus tejidos para investigación médica."
  Interventions: Other: NCI-developed educational materials

INTERVENTIONS:
Other: TBCCN-developed educational materials — Participants will be asked to view the educational materials developed by TBCCN, in either English or Spanish depending on the RCT in which they are enrolled. These materials include a DVD and a booklet that were developed to enhance community members' understanding and awareness of biospecimen collection and biobanking from healthy individuals.
  Arms: TBCCN-developed educational materials
Other: NCI-developed educational materials — Participants will be asked to view the English biobanking educational Brochure entitled "Providing your Tissue for Research: What you need to Know", or Spanish brochure entitled "Lo que usted debe saber antes de dar sus tejidos para investigación médica."
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate English and Spanish language educational materials that inform the community about a type of cancer research that involves the collection, storage, and processing of biospecimens. Part A of this study involved creating surveys about biospecimen donation and research. Now, a randomized controlled trial (RCT) will begin to evaluate education materials about biospecimen donation and research.

Phase II consists of two independent randomized controlled trials. Each trial is being conducted independently to test English and Spanish language materials (75 subjects each).

DETAILED DESCRIPTION:
The project addresses gaps in information by developing and validating English and Spanish language instruments to measure knowledge of and attitudes towards biospecimen donation and banking, as well as intention to donate biospecimens to a biobank (Part A). Once developed, the instruments will be used to evaluate biobanking educational priming tools by conducting two independent RCTs. Wherein English educational materials will be tested with 75 participants recruited from an urban clinic, and Spanish educational materials will be tested with 75 participant recruited form a rural community health center network. For each RCT following baseline assessment, participants will be randomized to either: 1) educational priming tools (DVD and booklet) developed by the Tampa Bay Community Cancer Network (TBCCN); or 2) an NCI-developed brochure entitled "Providing Your Tissue for Research: What You Need to Know." Seven to 28 days later participants will be given a telephone follow up interview.

ELIGIBILITY:
English Language RCT Inclusion Criteria:

* scheduled for an appointment at Lifetime Cancer Screening (LCS)
* able to read and speak English
* able to provide informed consent

Spanish Language RCT Inclusion Criteria:

* receiving care at a participating clinic from the Suncoast Community Health Centers network
* able to read and speak Spanish
* able to provide informed consent

Exclusion Criteria:

* previously diagnosed with cancer
* previously participated in a biobank
* participated in another TBCCN-related study entitled "community perceptions on biobanking"

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2010-09-27 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
BANKS-Knowledge Scale | Average of 28 days
  Administered at baseline and between 7 and 28 days after enrollment. Description: A validated 16-item questionnaire measuring knowledge about biobanking.
BANKS-Attitudes Scale | Average of 28 days
  Administered at baseline and between 7 and 28 days after enrollment. Description: A validated 15-item questionnaire measuring attitudes toward biobanking.
BANKS-Self-Efficacy Scale | Average of 28 days
  Administered at baseline and between 7 and 28 days after enrollment. Description: A validated 12-item questionnaire measuring self-efficacy in regards to donating a biospecimen to a biobank.
BANKS-Intentions | Average of 28 days
  Administered at baseline. Description: A single item measuring intentions to donate a biospecimen to a biobank.
Decisional Self-Efficacy | Average of 28 days
  Administered at follow-up (between 7 and 28 days after enrollment). Description: A validated 11-item questionnaire measuring participant's confidence in making a decision about donating a biospecimen (O'Connor M.A. Decision Self-efficacy Scale. 1995; www.ohri.ca/decisionaid).

SECONDARY OUTCOMES:
BANKS-Trust Scale | Average of 28 days
  Administered at baseline and between 7 and 28 days after enrollment. Description: A validated 10-item questionnaire measuring trust related to organizations, facilities, and people that may be involved in research.

CONTACTS AND LOCATIONS:
Overall Officials: Clement Gwede, PhD, MPH, RN, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States